CLINICAL TRIAL: NCT02978014
Title: A Randomised Controlled Phase II Trial Assessing Post-Operative Use of ProSpare, a Rectal Obturator in Prostate Cancer Radiotherapy
Brief Title: A Trial Assessing Post-Operative Use of ProSpare, a Rectal Obturator in Prostate Cancer Radiotherapy
Acronym: POPS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCR 4359
Record Dates: First submitted 2016-11-25; First posted 2016-11-30 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Cancer
Keywords: Prostate; Radiotherapy; Obturator; Toxicity; Bowel; Urinary; Sexual; PROM; EPIC
MeSH Terms: conditions — Neoplasms; Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ProSpare Arm (Experimental): ProSpare (obturator) image guided IMRT (i.e. radiotherapy administered to patients with the ProSpare device inserted in the rectum)
  Interventions: Device: ProSpare
- Non-ProSpare Arm (No Intervention): Standard of Care (non-obturator) image guided IMRT (i.e. radiotherapy administered to patients without the ProSpare device inserted in the rectum)

INTERVENTIONS:
Device: ProSpare — A novel rectal obturator (ProSpare) acting as a non-invasive daily on-line image guided tool, a rectal spacer and a prostate bed stabiliser
  Other Names: Rectal obturator
  Arms: ProSpare Arm

SUMMARY:
A two-arm randomised controlled trial in patients receiving post-prostatectomy radiotherapy in the adjuvant or salvage setting, with patients randomised to receive daily ProSpare (obturator) guided IMRT or Centre standard (non-obturator) guided IMRT.

DETAILED DESCRIPTION:
Surgery to remove the prostate gland is one of the ways of treating prostate cancer. Some patients receive radiotherapy after surgery if the cancer may not have been completely removed. Radiotherapy to the area where the prostate was can cause side effects, which can cause bowel and bladder symptoms as well as reducing sexual function.

Radiotherapy alone is also a standard treatment for prostate cancer. At the Royal Marsden Hospital and Institute of Cancer Research the investigators have designed and patented a device called ProSpare to improve the accuracy of radiotherapy. The device has already been developed and tested in over 80 patients having prostate radiotherapy and was well tolerated. Treatment accuracy was improved and the radiation dose to the rectum was reduced. Patients have given very valuable feedback and comments about ProSpare's design and use, which the investigators have incorporated in the final design. It is now important to test ProSpare in a multi-centre randomised controlled trial. The investigators aim to determine whether ProSpare will reduce the side effects reported by patients having radiotherapy after prostatectomy.

The ProSpare device is inserted by the patient into the rectum for each daily radiotherapy treatment. The disposable device stays in place for about 15 minutes each day. The curve in the device is designed to follow the shape of the rectum and it stays in the correct place by securely locating in the anal sphincter. ProSpare contains small "markers" - steel ball bearings - which can be "seen" on the standard scans taken before a radiotherapy treatment. Treatment is adjusted before each daily treatment to account for patient movement and radiotherapy set-up variation. As a result, treatment is more accurate than using the standard methods of radiotherapy localisation. This means the radiotherapy "safety margins" which are placed around the prostate bed can be reduced. The dose to the rectum and bladder as well as the structures that are associated with erectile function will be reduced. This may lead to an improvement in the side effects caused by radiotherapy.

Other ways to identify the treatment target area for such image guided radiotherapy (IGRT) includes the insertion of fiducial markers - usually in the form of gold seeds into the prostate or prostate bed. This has become standard practice in some radiotherapy centres for prostate radiotherapy but is technically complex for prostate bed radiotherapy and not routinely used. ProSpare has the additional advantage of being non-invasive and without the risk of infection associated with fiducial insertion.

Patients will be randomly selected to either have standard treatment or use ProSpare daily with adjusted set-up margins. During and after treatment, patients will be asked questions and given questionnaires to complete, asking about bowel, urinary and sexual function. The investigators will look at the results in each group and see if treatment with ProSpare has a benefit in improving the side effects from radiotherapy. If a benefit is seen, the aim will be for ProSpare guided radiotherapy to become part of the standard treatment for prostate bed radiotherapy nationally and internationally.

ELIGIBILITY:
Inclusion criteria:

1. Patient has undergone radical prostatectomy
2. Histologically confirmed prostatic cancer
3. Patient due to receive post-operative prostate bed radiotherapy either in the adjuvant or salvage* setting
4. WHO performance status 0-1 at randomization
5. Age > 18 years
6. Written informed consent
7. Able to independently complete patient questionnaires

Exclusion Criteria:

1. Lymph node or distant metastases from prostate cancer
2. Prior pelvic radiotherapy
3. Previous invasive cancer in the past 3 years, with the exception of non-melanoma skin cancer
4. Symptomatic haemorrhoids or other anal conditions which affect adequate insertion and retention of the rectal obturator
5. Planned chemotherapy within 2 months of completion of adjuvant or salvage radiotherapy
6. Musculoskeletal conditions which limit flexibility or mobility and will make patient self insertion of ProSpare™ difficult
7. Comorbid conditions likely to impact on advisability of prostate bed radiotherapy (e.g. inflammatory bowel disease, previous colorectal surgery, significant bladder instability or urinary incontinence)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Estimated)
Dates: Start 2017-02-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
EPIC Bowel Scores for Bowel, Urinary and Sexual domains | Two years
  Difference between groups in EPIC scores

SECONDARY OUTCOMES:
Quality of Life measures | Two and Five years
  Six Patient Reported Outcome Measure (PROM) questionnaires
Dosimetric analysis | Two years
  Analysis of dose/toxicity axis

CONTACTS AND LOCATIONS:
Overall Officials: Dr Julia Murray, Principal Investigator — Royal Marsden Hospital / Institute of Cancer Research
Locations (10):
- United Kingdom (10):
  - Beacon Centre, Musgrove Park Hospital, Taunton, Somerset
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - Cambridge University Hospitals, Cambridge
  - Royal Surrey County Hospital NHS Foundation Trust, Guildford
  - East Suffolk and North Essex NHS Trust, Ipswich
  - University College London Hospitals NHS Foundation Trust, London
  - Royal Free Hampstead NHS Trust, London
  - The Royal Marsden NHSFT, London
  - East and North Hertfordshire NHS Trust, Mount Vernon Cancer Centre, Middlesex
  - Norfolk and Norwich University Hospital NHSFT, Norwich

IPD SHARING:
Plan to Share IPD: No
We have not made a plan to share IPD at this stage but will finalise this following the first meeting of the Trial Management Group in Spring 2017